CLINICAL TRIAL: NCT02633124
Title: Preventing Catheter-related Bacteremia When Administering Injectable Medications in Premature Infants: Randomized Controlled Multicenter Study of Edelvaiss Multiline NEO Device
Brief Title: Preventing Catheter-related Bacteremia When Administering Injectable Medications in Premature Infants.
Acronym: MultilineNEO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2014_67; 2015-A00585-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Bacteremia; Infant, Very Low Birth Weight
Keywords: Premature infants; Catheter-related bacteremia; Infusion device; Neonatal intensive care; Central Venous Catheter; Drug Infusion Systems
MeSH Terms: conditions — Bacteremia; Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edelvaiss Multiline NEO (Experimental): The Edelvaiss Multiline NEO design allows to position the access to the infusion line outside of the incubator, without increasing the residual volume and this device has been validated by the manufacturer as part of CE marking for a period of 21 days.
  Interventions: Device: Edelvaiss Multiline NEO
- Standard Infusion Set (Other): The infusion set used for the standard group is the infusion set usually used.
  Interventions: Device: Standard Infusion Set

INTERVENTIONS:
Device: Edelvaiss Multiline NEO — Use of Edelvaiss Multiline NEO to infuse the parenteral nutrition and drugs during the study period
  Arms: Edelvaiss Multiline NEO
Device: Standard Infusion Set — Use of Standard Infusion Set to infuse the parenteral nutrition and drugs during the study period
  Arms: Standard Infusion Set

SUMMARY:
This study evaluates the potential interest of a new multi-lumen infusion access device (Edelvaiss® Multiline NEO) in the prevention of catheter-related bacteremia when administering injectable drugs in premature infants. This device will be compared to the standard infusion set of each center.

DETAILED DESCRIPTION:
Edelvaiss® Multiline NEO is a multi-lumen infusion access device, adapted to the neonatal population. It has five ports connected to five lumens separated in a single tube of 90 cm, combined with a small single tube called annex port. Four ports numbered 1 to 4 are connected to four peripheral lumens (residual volume per lumen: 0.6 mL). The fifth port, called central access (indicated by the HF icon (High Flow)), is reserved to the administration of parenteral nutrition. It is connected to the central lumen (residual volume: 4.5 mL). The sixth port on the annex way allows an administration closer to the infant (residual volume: 0.40 mL). It is thus reserved for emergencies and direct intravenous injections.

The innovative technological design of Edelvaiss® Multiline NEO device should enable secure administration of injectable drugs by preventing variations in drug mass flow rate and the occurrence of drug incompatibilities. This device would reduce the number of perfusion incidents and therefore, the frequency of manipulations of infusion lines within the incubator, direct source of occurrence of bacteremia.

Moreover, its main interest lies in neonatology in the possibility of being positioned outside of the incubator and to have a lifetime of 21 days, contributing to the prevention of catheter-related bacteremia. All manipulations are therefore made outside the incubator at the room temperature and the relative humidity, and at a distance from the device/catheter junction.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational ages between 24 and 29 weeks.
* Infants carrying a single-lumen central venous catheter.
* Obtaining the informed parental consent.

Exclusion Criteria:

* Infants carrying a multi-lumen central venous catheter.
* Infants carrying a umbilical venous catheter.
* Infants carrying two central venous catheters.
* Refusal of informed parental consent.

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Measure of incidence density (ID) of catheter-related bacteremia (CRB) | Through an average of 30 days
  Catheter-related bacteremia (CRB) are the most frequent nosocomial infections in Neonatal Intensive Care Unit (NICU) patients. Nosocomial CRB in the NICU contribute significantly to hospital morbidity as well as to increased costs due to prolonged hospitalization.
  The main objective is to assess the interest of the Multiline NEO in preventing CRB when administering injectable medications in NICU patients. It is whether the Multiline NEO device reduces the risk of CRB in premature infants hospitalized in NICU.
  Measure of ID of CRB as criteria of Neocat Network during central venous catheterization in the patient.

SECONDARY OUTCOMES:
Measure of ID of occlusion of components of the infusion system | Through an average of 30 days
  Measure of ID of occlusion of components of the infusion system is determined on the period of central venous catheterization in the patient.
Number of septic shock | Through an average of 30 days
  The number of septic shock defined by the use of vasoactive drugs during central venous catheterization in the patient.
Total duration of oxygen therapy | Through an average of 30 days
  Total duration of oxygen therapy is determined from the inclusion of the patient in the study until the end of his hospitalization.
Total duration of mechanical ventilation | Through an average of 30 days
  Total duration of mechanical ventilation is determined from the inclusion of the patient in the study until the end of his hospitalization.
Total duration of parenteral nutrition | Through an average of 30 days
  Total duration of parenteral nutrition is determined from the inclusion of the patient in the study until the end of his hospitalization.
Number of bronchopulmonary dysplasia | Through an average of 30 days
  Number of bronchopulmonary dysplasia defined by the Walsh test is determined from the inclusion of the patient in the study until the end of his hospitalization.
Cost of care for patients | Through an average of 30 days
  Cost of care for patients includes :
  * cost of components of the infusion lines, including their replacement,
  * cost of nursing time dedicated to handling lines,
  * cost of identifying a CRB,
  * cost of hospital stay. Cost of care for a patient is calculated from the inclusion of the patient in the study until the end of his hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Storme, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Chu Amiens Picardie, Amiens
  - Hôpital Côte de Nacre - CHU de Caen, Caen
  - Hôpital Jeanne de Flandre - CHRU de Lille, Lille
  - Hôpital Charles Nicolle - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mahieu LM, De Dooy JJ, Lenaerts AE, Ieven MM, De Muynck AO. Catheter manipulations and the risk of catheter-associated bloodstream infection in neonatal intensive care unit patients. J Hosp Infect. 2001 May;48(1):20-6. doi: 10.1053/jhin.2000.0930. PMID 11358467
- [Result] Erdei C, McAvoy LL, Gupta M, Pereira S, McGowan EC. Is zero central line-associated bloodstream infection rate sustainable? A 5-year perspective. Pediatrics. 2015 Jun;135(6):e1485-93. doi: 10.1542/peds.2014-2523. Epub 2015 May 18. PMID 25986020
- [Derived] Maiguy-Foinard A, Decaudin B, Tourneux P, Guillois B, Blanc T, Galene-Gromez S, Masse M, Odou P, Denies F, Dervaux B, Duhamel A, Storme L. Effect of multi-lumen perfusion line on catheter-related bacteremia in premature infants: study protocol for a cluster-randomized crossover trial. Trials. 2019 Feb 11;20(1):115. doi: 10.1186/s13063-019-3218-6. PMID 30744679
- See also: Website of the Multiline NEO manufacturer (Doran International) — http://www.doran-int.com/